CLINICAL TRIAL: NCT06693609
Title: A Phase 2a, Exploratory, Randomized, Double-Blind, Placebo-Controlled Trial of the Safety, Tolerability, and Efficacy of EMP-01 in Adult Participants With Social Anxiety Disorder
Brief Title: Exploratory Safety and Efficacy of EMP-01 in Social Anxiety Disorder
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: atai Therapeutics, Inc. (Industry)
Collaborators: EmpathBio, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMP-01-201
Record Dates: First submitted 2024-11-12; First posted 2024-11-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-04

CONDITIONS: Social Anxiety Disorder
Keywords: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Intervention Model Description: A Phase 2a, Exploratory, Randomized, Double-Blind, Placebo-Controlled Trial of the Safety, Tolerability, and Efficacy of EMP-01 in Adult Participants with Social Anxiety Disorder
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EMP-01 (Experimental)
  Interventions: Drug: EMP-01
- EMP-01 Placebo (Placebo Comparator)
  Interventions: Drug: EMP-01 Placebo

INTERVENTIONS:
Drug: EMP-01 — EMP-01 capsules
  Arms: EMP-01
Drug: EMP-01 Placebo — EMP-01 placebo capsules
  Arms: EMP-01 Placebo

SUMMARY:
This Phase 2 study (protocol number EMP-01-201) will determine the safety and tolerability of a short-term treatment with an oral dosage form of EMP-01 in adult participants with social anxiety disorder (SAD) and will assess exploratory efficacy of repeated doses of EMP-01 versus placebo.

DETAILED DESCRIPTION:
This Phase 2, exploratory, multi-center, double-blind, randomized, placebo-controlled trial will enroll approximately 60 adult participants with SAD, randomized 1:1 to receive a total of 2 double-blind administrations of EMP-01 or placebo with a 4-week interval between each administration during the placebo-controlled treatment period. All participants will have their symptoms monitored for 6 weeks until the conclusion of the study. While the primary objective of the study is to assess the safety and tolerability of EMP-01 in participants with SAD, the secondary objective is to estimate any improvement in social anxiety symptoms of participants compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

Eligibility will be assessed at Screening and will be reconfirmed on Day -1 (Baseline) based on available information, before randomization on the following day (Day 1).

Participants must meet all of the following criteria to be enrolled in this study:

Age

1. Participants must be between 18 and 65 years of age, inclusive, at the time of signing the ICF.

   Disease Characteristics
2. Has a current diagnosis of SAD, as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition Text Revision (DSM-5-TR), which is not better attributable to another psychiatric condition or to a medical condition. The diagnosis will be confirmed by the Mini-International Neuropsychiatric Interview (MINI).
3. Clinician-administered LSAS total score ≥ 70 at Screening and Day -1.
4. Clinician Global Impressions - Severity (CGI-S) score ≥ 4 at Screening and Day-1.

   Weight
5. Body mass index (BMI) within the range 20-34 kg/m2 (inclusive) at Screening.
6. Able (in the investigator's opinion) to comprehend and be willing to sign an ICF, to abide by the study restrictions, and to attend all study visits.

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from this study:

Medical Conditions

1. Has a current or prior DSM-5-TR diagnosis of a schizophrenia spectrum and other psychotic disorder, substance/medication-induced psychotic disorder, bipolar and related disorder, or any disorder with psychotic features (including MDD with psychotic features), as assessed by medical history and a structured clinical interview (MINI).
2. Has a current or prior DSM-5-TR diagnosis of a neurocognitive disorder, intellectual disorder, dissociative disorder, disruptive/impulse-control/conduct disorder, autism spectrum disorder (level 2 or 3), or cluster A and B personality disorder, as assessed by medical history and a structured clinical interview (MINI). Inclusion of individuals with a diagnosis of autism spectrum disorder level 1 may be considered at the discretion of the investigator if the participant no longer meets criteria for the condition and current functioning and/or subthreshold symptoms will not interfere with treatment or compliance in the study.
3. Has a current DMS-5-TR diagnosis of SAD performance only sub-type, PTSD, acute stress disorder, anorexia nervosa, bulimia nervosa, or any other co-morbid psychiatric condition that dominates the clinical presentation and would interfere with experimental treatment.
4. Has a current DMS-5-TR disorder, other than SAD, which is the primary focus of treatment. Note that participants with concurrent GAD are eligible for the study, provided that GAD is not the primary diagnosis. Participants with attention deficit hyperactivity disorder (ADHD) are eligible for the study, provided that they do not require pharmacological treatment for the condition AND if ADHD is not the primary diagnosis.
5. Has severe current depression, as measured by a total score ≥ 16 on the QIDS-SR-16.
6. Has a history of moderate or severe alcohol or cannabis use disorder within 1 year before Screening. Has any severity (including mild) of other substance use disorder (drug) within 1 year before Screening, as confirmed by the MINI.
7. Has had suicidal ideation with some intent to act within 6 months before Screening or a history of suicidal behavior within the past 1 year before Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-02-04 (Estimated); Study Completion 2026-02-04 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events, adverse events of special interest and serious adverse events. | Day 1 to EOS [Day 43]
  Assess the safety and tolerability of EMP-01 compared with placebo (PBO) in participants with SAD.
Incidence of clinically significant abnormalities in physical examinations, vital signs, electrocardiogram parameters, and safety laboratory results. | Day 1 [post-dose] to Day 57
  Assess the safety of EMP-01 compared with placebo (PBO) in participants with SAD.
Columbia-Suicide Severity Rating Scale (C-SSRS) Score | Baseline to Day 57
  Assess the safety of EMP-01 compared with placebo (PBO) in participants with SAD.

SECONDARY OUTCOMES:
Liebowitz Social Anxiety Scale (LSAS) | Baseline to EOS [Day 43]
  Change from Baseline in the Liebowitz Social Anxiety Scale (LSAS) total score at Day 43 to evaluate the treatment difference in EMP-01 compared with PBO in improving social anxiety symptoms in participants with SAD 6 weeks after initiating treatment.

CONTACTS AND LOCATIONS:
Locations (7):
- United Kingdom (7):
  - MAC Clinical Research - South Staffordshire, Bridgetown, Cannock, Staffordshire
  - MAC Clinical Research - Greater Manchester, Manchester, Greater Manchester
  - MAC Clinical Research - Lancashire, Blackpool, Lancashire
  - MAC Clinical Research - Merseyside, Liverpool, Merseyside
  - MAC Clinical Research - South Yorkshire, Tankersley, South Yorkshire
  - MAC Clinical Research - Teesside, Thornaby, Stockton-on-Tees
  - MAC Clinical Research Centre, West Yorkshire, Leeds

IPD SHARING:
Plan to Share IPD: No